CLINICAL TRIAL: NCT03914677
Title: Pilot Study of Mecamylamine for Autonomic Dysreflexia Prophylaxis
Brief Title: Mecamylamine for Autonomic Dysreflexia Prophylaxis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Edward Nieshoff, MD, Principal Investigator, Wayne State University
Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 080518MP2F
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; autonomic dysreflexia; mecamylamine
MeSH Terms: conditions — Spinal Cord Injuries; Autonomic Dysreflexia | interventions — Mecamylamine

STUDY DESIGN:
Intervention Model Description: dose-escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Mecamylamine Oral Tablet (Experimental): Initial dose - mecamylamine 2.5 mg tablet po 3 hours prior to provocative testing; subsequent dose escalations as needed, to 5 mg and then 7.5 mg, using the same testing methodology.
  Interventions: Drug: Mecamylamine Oral Tablet

INTERVENTIONS:
Drug: Mecamylamine Oral Tablet — nicotinic antagonist (ganglionic blocker)
  Other Names: Vecamyl

SUMMARY:
This is a preliminary study of the antihypertensive drug mecamylamine, used in the specific circumstance of hypertension caused by autonomic dysreflexia (AD), a condition that affects people with spinal cord injury (SCI). Initially, mild sensory stimulation of subjects' legs is used to intentionally provoke AD, as reflected by blood pressure elevation during such stimulation. In subsequent testing sessions, mecamylamine is given prior to sensory stimulation, to show the effect of the drug on preventing these AD-related blood pressure elevations.

DETAILED DESCRIPTION:
In this one year pilot study we will enroll 3-5 people with SCI, and aim to develop a simple, convenient BP cuff method to elicit AD (i.e., using a BP cuff applied to the leg as a mild noxious stimulus), and then use that method to preliminarily evaluate the effects of the antihypertensive drug mecamylamine on AD. Study participants will complete up to 5 research visits, will undergo AD provocation using the leg cuff protocol, and will receive escalating doses of mecamylamine, as needed and tolerated, in order to prevent AD:

After signing the informed consent form, at visit 1, subjects will complete an interview to evaluate past medical history, an autonomic dysfunction questionnaire, a physical examination (including an autonomic assessment and specialty SCI exam), vital signs measurement, and baseline testing of the electrical activity of the heart (electrocardiography or ECG testing).

At visit 2, subjects will complete a preparation procedure including: baseline vital signs measurement, an interview to document all medications and/or supplements taken in the prior 24 hours, confirmation of completed bladder/bowel evacuation before the visit, confirmation of no significant illness/injury since last visit, and documentation of any meals before the visit. Next, the subject will be connected to an ECG monitor and a (second) BP cuff will be applied to the arm (for measuring BP response to the leg cuff procedure). With the ECG and arm cuff in place, s/he will undergo the AD provocation procedure: The BP cuff placed around the leg just below the knee will be inflated for up to 10 minutes, as a means of providing sensory stimulation to elicit AD. BP will be measured using the arm cuff every 2 minutes during the leg cuff inflation, and periodically after the leg cuff is deflated, until BP and heart rate are back to baseline values. Physical manifestations and symptoms of AD will be recorded during the period of leg cuff inflation and thereafter, throughout recovery. This BP cuff protocol will be repeated twice during the same visit, with trials separated by a 30-minute recovery period. The leg cuff will be deflated immediately if the blood pressure-measuring cuff shows that systolic BP exceeds 180 mmHg, diastolic BP exceeds 100 mmHg, heart rate is less than 40 or greater than 100 beats per minute, adverse ECG changes are evident, or symptoms are unacceptable to the subject. An established safety plan will be followed in the event of a significant adverse reaction to the leg compression or study drug. If the leg cuff inflation fails to elicit AD, then the subject will be dropped from the study.

At visit 3, a similar visit preparation procedure will be completed as in visit 2. Three hours prior to AD provocation testing with the leg cuff, subjects will receive 2.5 mg of mecamylamine in tablet form, to try to prevent AD. Physical manifestations and symptoms of AD will be recorded during the period of cuff inflation and thereafter, throughout recovery. The leg cuff will be deflated after 10 minutes, or immediately as appropriate according to the same criteria as listed for visit 2. After a 30-minute recovery, the leg cuff inflation will be repeated once during the same session, to confirm whether or not 2.5 mg of mecamylamine eliminates AD, or at least reduces the associated BP elevation, as well as the other manifestations and symptoms. If the dose of 2.5 mg mecamylamine is effective, the subject will not be asked to return for testing with a higher dose and study participation will end with visit 3. If either trial of leg cuff inflation still elicits AD despite premedication with 2.5 mg mecamylamine, then s/he will be scheduled to come back for visit 4.

At visit 4, the visit preparation will be completed as in visits 2 and 3. Three hours prior to testing with the AD provocation procedure, 5 mg of mecamylamine will be given to the participant to try to prevent AD, since the lower dose failed to do so. The same procedures described above for visit 3 will be followed; subjects will again undergo 2 trials of AD provocation with the leg squeezing procedure. If both are successful (i.e., no AD is observed), the subject's participation in the study will end. If, despite premedication with mecamylamine 5 mg, the subject still experiences AD, then s/he will be asked to return for visit 5.

At visit 5, all the procedures as in visit 4 will be repeated, except that subjects will receive 7.5 mg of mecamylamine. Regardless if the medication does not prevent AD, subjects will not be scheduled to come for a follow up, as no further dose escalation will be attempted.

If at visit 3, 4, or 5 a subject experiences symptomatic low blood pressure after taking mecamylamine (manifest as dizziness, lightheadedness, or change in vision; this is considered unlikely based on the published literature), s/he will be asked to drink several glasses of cold water, and possibly to lay down for up to 30 minutes to try to alleviate those symptoms. In the event symptomatic low blood pressure persists, the subject will be given 10 mg of midodrine, a medication to elevate blood pressure. Midodrine would be expected to promptly (in less than an hour) elevate blood pressure and alleviate those symptoms. Upon adequate elevation of blood pressure to cause resolution of the symptoms, the subject will be discharged from the study, because of the adverse effect of mecamylamine. If the midodrine 10 mg fails to resolve symptomatic low blood pressure, then further evaluation and treatment will be provided as appropriate (e.g., intravenous fluids). The latter scenario is considered to be extremely unlikely.

note - visits will be separated by no more than one month

ELIGIBILITY:
Inclusion Criteria:

* chronic (>1 year) SCI at T6 or above, American Spinal Injury Association grade A, B, or C
* negative serum pregnancy test for females

Exclusion Criteria:

* history of arrhythmia, cardiovascular disease, cerebral aneurysm
* contraindications to use of mecamylamine or midodrine (pregnancy, nursing, glaucoma, kidney disease, pyloric stenosis, arteriosclerosis, or concurrent use of a sulfonamide antibiotic)
* dependence on reflex voiding for bladder management (mecamylamine may cause urinary retention)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2020-03-17 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
change in systolic blood pressure | 10 minutes (following initiation of sensory stimulation)
  difference in systolic blood pressure during leg cuff inflation vs during unstimulated baseline
change in heart rate | 10 minutes (following initiation of sensory stimulation)
  difference in heart rate during leg cuff inflation vs during unstimulated baseline

SECONDARY OUTCOMES:
signs and symptoms of autonomic dysreflexia | 10 minutes (following initiation of sensory stimulation)
  piloerection, diaphoresis, headache

CONTACTS AND LOCATIONS:
Overall Officials: EDWARD C NIESHOFF, MD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available for all primary and secondary outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 6 months following completion of the study through 5 years after completion.
Access Criteria: Data access requests will be reviewed by the Research Director of the sponsoring Wayne State University Department of Physical Medicine and Rehabilitation. Data will be made available to researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Braddom RL, Johnson EW. Mecamylamine in control of hyperreflexia. Arch Phys Med Rehabil. 1969 Aug;50(8):448-53 passim. No abstract available. PMID 5806088
- [Background] Braddom RL, Rocco JF. Autonomic dysreflexia. A survey of current treatment. Am J Phys Med Rehabil. 1991 Oct;70(5):234-41. PMID 1910647
- [Background] Eldahan KC, Rabchevsky AG. Autonomic dysreflexia after spinal cord injury: Systemic pathophysiology and methods of management. Auton Neurosci. 2018 Jan;209:59-70. doi: 10.1016/j.autneu.2017.05.002. Epub 2017 May 8. PMID 28506502
- [Background] Groothuis JT, Rongen GA, Deinum J, Pickkers P, Danser AH, Geurts AC, Smits P, Hopman MT. Sympathetic nonadrenergic transmission contributes to autonomic dysreflexia in spinal cord-injured individuals. Hypertension. 2010 Mar;55(3):636-43. doi: 10.1161/HYPERTENSIONAHA.109.147330. Epub 2010 Jan 25. PMID 20100992